CLINICAL TRIAL: NCT06692257
Title: Orofacial Functions With Emphasis on Breathing and Chewing Patterns in Individuals With and Without Molar Incisor Hypomineralization: Observational Study Protocol
Brief Title: Orofacial Functions in Individuals With and Without Molar Incisor Hypomineralization
Status: Not yet recruiting | Type: Observational
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Principal Investigator, University of Nove de Julho
Other Study IDs: Orofacial functions
Record Dates: First submitted 2024-11-14; First posted 2024-11-18 (Actual); Last update posted 2024-11-18 (Actual); Status verified 2024-11

CONDITIONS: Molar Hypomineralization, Incisor
MeSH Terms: conditions — Molar Hypomineralization | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Individuals without MIH: All permanent molars without indices compatible with MIH
  Interventions: Behavioral: Observation
- Individuals with MIH: At least one permanent molar with indices compatible with MIH (code 2, 21, 22 and 3 - Ghanim criteria)
  Interventions: Behavioral: Observation

INTERVENTIONS:
Behavioral: Observation — To perform a comparative analysis of orofacial functions with an emphasis on breathing and chewing patterns in individuals with and without MIH.

SUMMARY:
Molar incisor hypomineralization (MIH) is a qualitative developmental defect of the enamel with a complex, multifactorial nature and a significant genetic component that predominantly affects the permanent first molars and, occasionally, the permanent incisors. Individuals with MIH have a compromised stomatognathic system manifested by muscle hyperactivity under postural and dynamic conditions. However, there is a gap in knowledge on the specific functional abnormalities that these individuals experience. Early identification and intervention, with a focus on the prevention of orofacial dysfunctions and deviations in facial growth and development, are aspects of the utmost importance. Therefore, the aim of the proposed study is to perform a comparative analysis of orofacial functions with an emphasis on breathing and chewing patterns in individuals with and without MIH. Methods and Analysis: Assessments will be performed using the Nordic Orofacial Test - Screening (NOT-S). Descriptive statistics will be performed and comparisons will be made using the chi-square test, adopting a 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* Children 6 to 12 years of age with a complete mixed dentition with all first molars present and in occlusion;
* Having all first molars erupted, without caries or previous treatment;
* Inclusion criteria for the MIH group: at least one permanent molar with indices compatible with MIH (code 2, 21, 22 and 3 - Ghanim criteria).

Exclusion Criteria:

* Children with amelogenesis and dentinogenesis imperfecta;
* Children undergoing orthodontic treatment;
* Children with a genetic syndrome;
* Children with the premature loss of deciduous teeth;
* Children with acute respiratory problems;
* Children in treatment.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The study will be conducted with children 6 to 12 years of age enrolled at the pediatric dentistry clinic of Nove de Julho University. The participants will be assessed in a single session during a visit to the clinic. All assessments will be performed by the same researcher.
Sampling Method: Probability Sample
Enrollment: 56 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of orofacial function (NOT-S) - (score from 0 to 12) | Baseline
  The following functions are addressed during the interview: (I) sensory function, (II) breathing, (III) habits, (IV) chewing and swallowing, (V) drooling and (VI) dryness of the mouth. The following functions are evaluated during the physical examination: (1) face at rest, (2) nose breathing, (3) facial expression, (4) masticatory muscle and jaw function, (5) oral motor function and (6) speech. For the evaluation of orofacial dysfunction during the clinical examination, the participants will be asked to perform tasks for each item in accordance with the illustrated manual. Each item has criteria for the respective function. A "YES" response or task the meets the criteria for compromised function will be scored 1 point, indicating dysfunction in the respective domain. A "NO" response or task that does not meet the criteria will be scored zero. The total is the sum of the points of all domains and ranges from 0 to 12, with higher scores denoting greater orofacial disfunction.

SECONDARY OUTCOMES:
Assessment of hypersensitivity in teeth with MIH: Visual analog scale (VAS) | Baseline
  The Wong-Baker Faces Pain Scale was initially developed for children to facilitate communication about pain. This scale uses a set of faces that ranges from a smiling expression (without pain) to a crying expression (worse pain possible), enabling children to indicate the intensity of their pain in a visually understandable way. The scale is used with children three years of age and older, facilitating communication and improving the assessment so that the management of the pain can be addressed.
Schiff cold air sensitivity scale (SCASS) | Baseline
  The SCASS will be used to assess the child's response to the stimulus and will be scored as follows: 0 = no response to the stimulus; 1 = response to the stimulus, child considers stimulus painful; 2 = response to the stimulus, child moves away from stimulus; 3 = response to the stimulus, child moves away from the stimulus and asks for its immediate interruption.

REFERENCES:
- [Derived] Pernomiam FC, Mandetta ARH, Ribeiro CDPV, Camargo CCB, Romano IMF, Sobral APT, Mesquita-Ferrari RA, Fernandes KPS, Horliana ACRT, Duran CCG, Motta LJ, Bussadori SK. Orofacial functions with emphasis on breathing and chewing patterns in individuals with and without molar incisor hypomineralisation: observational study protocol conducted in a dental clinic in Brazil. BMJ Open. 2025 Jun 4;15(6):e101725. doi: 10.1136/bmjopen-2025-101725. PMID 40467310